CLINICAL TRIAL: NCT02409992
Title: Parent Training and Emotion Coaching for Children With Limited Prosocial Emotions
Acronym: HNC-EC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lynn Fainsilber Katz, Research Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000931
Record Dates: First submitted 2015-03-25; First posted 2015-04-07 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Oppositional Defiant Disorder
Keywords: Children with ODD and low prosocial emotions
MeSH Terms: conditions — Oppositional Defiant Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Training plus Emotion Coaching (Experimental): This intervention will combine a parent management training program called Helping the Noncompliant Child with elements of an Emotion Coaching parenting intervention.
  Interventions: Behavioral: Parent Training plus Emotion Coaching
- Parent Training Only (Active Comparator): This intervention will consist of a parent management training program called Helping the Noncompliant Child.
  Interventions: Behavioral: Parent Training only

INTERVENTIONS:
Behavioral: Parent Training plus Emotion Coaching — This intervention will combine a parent management training program called Helping the Noncompliant Child with elements of an Emotion Coaching parenting program.
  Arms: Parent Training plus Emotion Coaching
Behavioral: Parent Training only — This intervention will consist of a parent management training program called Helping the Noncompliant Child.
  Arms: Parent Training Only

SUMMARY:
The proposed research will focus on the development of a brief emotion-coaching (EC) parenting program (which directly targets child emotion awareness/recognition and affective empathy), that will be combined with a well-established parent management training program (Helping the Noncompliant Child; HNC) for treating oppositional defiant disorder (ODD) in children who also have limited prosocial emotions (e.g., lack of guilt and empathy, callous use of others).

ELIGIBILITY:
Inclusion Criteria:

* Child with oppositional defiant disorder and low prosocial emotions

Exclusion Criteria:

* Unable to speak/understand English
* Significant developmental delay or autism spectrum disorder

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory - intensity score | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Child conduct problems at baseline, mid-treatment and post-treatment
Early Childhood Inventory-4 ODD scale | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Change in child conduct problems for children ages 3-5 at baseline, mid-treatment and post-treatment
Child Symptom Inventory-IV | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Child conduct problems for children ages 6-7 at baseline, mid-treatment and post-treatment
Behavioral Coding System - percent child inappropriate behaviors | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Child inappropriate behaviors at baseline, mid-treatment and post-treatment
Behavioral Coding System percent child compliance | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Child compliance at baseline, mid-treatment and post-treatment

SECONDARY OUTCOMES:
Inventory of Callous-Unemotional Traits - preschool version - total score | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Callous-unemotional traits at baseline mid-treatment and post-treatment
A Developmental Neuropsychological Assessment (NEPSY-II) Affect Recognition Task - fear recognition | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Affect recognition at baseline, mid-treatment and post-treatment
NEPSY-II Affect Recognition Task - sadness recognition | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Affect recognition in baseline mid-treatment and post-treatment
Griffith Empathy Measure - empathy score | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Empathy at baseline and post-treatment
Behavioral coding of Zahn-Waxler empathy paradigm - amount of attention, affective response congruent with examiner, concern for others, disregard for others | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Empathy at baseline and post-treatment
Behavioral Coding System - positive attention rate per minute | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Parenting behavior - positive attention at baseline mid-treatment and post-treatment
Behavioral Coding System - total commands rate per minute | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Change in parenting behavior - commands at baseline mid-treatment and post-treatment
Parenting scale - overactivity | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Parenting at baseline mid-treatment and post-treatment
Parenting scale - laxness | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Parenting at baseline mid-treatment and post-treatment
Parent Meta-Emotion Interview emotion coaching scale | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Emotion coaching at baseline and post-treatment
Parenting Sense of Competence satisfaction scale | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Parenting satisfaction at baseline mid-treatment and post-treatment
Parenting Sense of Competence efficacy scale | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Parenting efficacy at baseline mid-treatment and post-treatment

OTHER OUTCOMES:
Difficulties with Emotion Regulation Scale - lack of awareness and limited access to emotion regulation strategies | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Maternal emotion regulation abilities at baseline mid-treatment and post-treatment
Beck Depression Inventory II | Participants will be followed for the duration of outpatient treatment, an expected average of 25 weeks
  Maternal depression at baseline and post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lynn F Katz, Ph.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States